CLINICAL TRIAL: NCT00062972
Title: Interventions to Improve Memory in Patients With Multiple Sclerosis
Brief Title: Improving Memory in Patients With Multiple Sclerosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated/withdrawn
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HD038107-01 (NIH)
Record Dates: First submitted 2003-06-18; First posted 2003-06-19 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2011-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cognitive Dysfunction; Treatment Interventions; Verbal memory deficits
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction | interventions — Donepezil; Glucose

INTERVENTIONS:
Drug: donepezil
Drug: glucose

SUMMARY:
People with multiple sclerosis (MS) suffer from cognitive and other brain problems. This study will examine the effectiveness of the drug donepezil and of sugar water for enhancing memory in individuals with MS. Donepezil (also known as Aricept) has been FDA approved for improving memory and learning in individuals with Alzheimer's disease.

DETAILED DESCRIPTION:
Cognitive dysfunction is one of the leading causes of disability in people with MS. Memory involving specific words (verbal memory) is particularly affected in individuals with MS. Attempts to rehabilitate cognitive dysfunction in MS have had only limited success.

This study will determine the efficacy of donepezil therapy and glucose administration for enhancing verbal memory functioning in individuals with MS. The study will also measure secondary outcomes assessing other areas of cognitive dysfunction (i.e., nonverbal memory, conceptual thinking, processing speed) which may improve with intervention.

Forty participants with MS will be randomly assigned to receive either donepezil or placebo for 24 weeks. Participants will complete memory and cognitive tests at the beginning and end of the 24 week period.

Twenty participants with MS will be randomly assigned to drink a beverage sweetened with either glucose or saccharin (placebo). Participants will then complete memory and other cognitive tests. Two weeks later, participants will drink a beverage sweetened with the alternative sweetener and again complete the memory and cognitive tests.

ELIGIBILITY:
Inclusion Criteria

* MS as defined by the Poser criteria
* Expanded Disability Status Scale (EDSS) score of 0 to 6.5
* Stable neurologic function for at least 30 days prior to study entry
* Agree to continue all current medications for study duration
* Rey Auditory Verbal Learning Test score in low normal range or below
* Mini-mental status exam score of 26 or higher
* Montgomery-Asberg Depression Scale scaled score of 14 or lower
* Fluent in English

Exclusion Criteria

* Use of anticholinergic or benzodiazepine medication
* Change in dosage of medications judged to have the potential to impact cognitive function (e.g., antispasticity medications) within 2 weeks of study entry
* Current alcohol or substance abuse
* History of neurological or major medical problem that has a known effect on cognitive functioning
* History of noncompliance
* Visual or upper extremity impairment which precludes ability to participate in cognitive assessment

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1999-09; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B. Krupp, MD, Principal Investigator — Department of Neurology, University Hospital Medical Center
Locations (1):
- University Hospital and Medical Center, Stony Brook, New York, United States

REFERENCES:
- [Background] Prosiegel M, Michael C. Neuropsychology and multiple sclerosis: diagnostic and rehabilitative approaches. J Neurol Sci. 1993 Apr;115 Suppl:S51-4. doi: 10.1016/0022-510x(93)90209-h. PMID 8340793
- [Background] Rudick R, Antel J, Confavreux C, Cutter G, Ellison G, Fischer J, Lublin F, Miller A, Petkau J, Rao S, Reingold S, Syndulko K, Thompson A, Wallenberg J, Weinshenker B, Willoughby E. Clinical outcomes assessment in multiple sclerosis. Ann Neurol. 1996 Sep;40(3):469-79. doi: 10.1002/ana.410400321. PMID 8797541
- [Background] Wild KV, Lezak MD,Whitman RH, Bourdette DN: Psychosocial impact of cognitive impairment in the multiple sclerosis patient. J Clin Exp Neuropsychology 415: 685-691, 1991
- [Background] Krupp LB, Sliwinski M, Masur DM, Friedberg F, Coyle PK. Cognitive functioning and depression in patients with chronic fatigue syndrome and multiple sclerosis. Arch Neurol. 1994 Jul;51(7):705-10. doi: 10.1001/archneur.1994.00540190089021. PMID 8018045
- [Background] Kujala P, Portin R, Revonsuo A, Ruutiainen J. Attention related performance in two cognitively different subgroups of patients with multiple sclerosis. J Neurol Neurosurg Psychiatry. 1995 Jul;59(1):77-82. doi: 10.1136/jnnp.59.1.77. PMID 7608714